CLINICAL TRIAL: NCT04366440
Title: De-Implementation of Unnecessary Surgical Antibiotic Prophylaxis in Children
Acronym: OPerAtiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201912100; 1R01HS026742-01A1 (AHRQ)
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Surgical Site Infection
Keywords: children; antimicrobial stewardship; post-operative antibiotic prophylaxis; Deimplementation
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: A stepped-wedge study design will be utilized. All sites will begin in the control intervention, order set review and modification. Sequentially, clusters of 3 hospitals will begin in the experimental intervention, order set review and modification plus facilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order set review and modification (Other): The antimicrobial stewardship program will review and change order sets of clean or clean-contaminated procedures to eliminate unnecessary post-operative antibiotics.
  Interventions: Other: Order set review and modification
- Order Set review and Modification plus facilitation (Other): The antimicrobial stewardship program will receive facilitation training to aid in reviewing and changing order sets of clean or clean-contaminated procedures to eliminate unnecessary post-operative antibiotics.
  Interventions: Behavioral: Order set review and modification with facilitation

INTERVENTIONS:
Behavioral: Order set review and modification with facilitation — The antimicrobial stewardship program will receive facilitation training to aid in reviewing and changing order sets of clean or clean-contaminated procedures to eliminate unnecessary post-operative antibiotics.
  Arms: Order Set review and Modification plus facilitation
Other: Order set review and modification — The antimicrobial stewardship program will work to eliminate unnecessary post-operative antibiotics by reviewing and changing order sets of clean or clean-contaminated procedures.
  Arms: Order set review and modification

SUMMARY:
The overall objective of this study is to identify the best strategy to eliminate unnecessary antibiotic use after surgery in pediatric surgical procedures considered low-risk for an SSI. Based on literature and our preliminary data suggesting surgeons will not fully accept standardized order sets based on current guidelines, the investigators hypothesize that order set modification combined with ASP facilitation will outperform standard order set modification alone in de-implementing unnecessary postoperative antibiotic use.

DETAILED DESCRIPTION:
Antibiotics have revolutionized healthcare allowing clinicians the ability to treat life-threatening infections and to prevent infections following life-saving surgery. Unfortunately, antibiotic overuse results in antibiotic resistant bacteria and unnecessary adverse events including Clostridioides difficile infections (CDI). Data demonstrate that antibiotic resistant bacteria and CDI annually kill up to 150,000 and 29,000 Americans, respectively. Surgical antibiotic prophylaxis is a common area for unnecessary antibiotic use among children. Recent CDC surgical site infection (SSI) guidelines and the AAP Choosing Wisely Campaign recommend no postoperative antibiotic prophylaxis for procedures considered low risk for an SSI.

In this study, our team will develop and test two theoretically informed strategies to eliminate ("de-implement") unnecessary postoperative antibiotic prophylaxis through the collaboration of surgeons and antimicrobial stewardship programs (ASPs). One promising strategy is the implementation of standard surgical order sets, which offer relative ease of implementation and a systematic approach across surgical subspecialties. While evidence suggests that order set standardization is a good approach, barriers to implementation are commonly noted, especially the lack of engagement with clinicians affected by change when initiating a new strategy. As such, complementary strategies are needed to extend the impact of order set standardization.

This study will be guided by the i-PARIHS framework (Integrated Framework for Promoting Action on Research Implementation in Health Services), an implementation science framework designed to guide implementation of evidence-based practices. This framework posits that successful implementation of evidence into practice is a function of the quality and type of evidence to be implemented, the characteristics of the context where the evidence will be implemented, and the means by which it is integrated or facilitated into practice. Four primary constructs comprise the i-PARIHS framework: the innovation, recipients, context, and facilitation. Innovation describes the evidence and knowledge regarding a particular issue, as well as the qualities of the evidence that may influence how it is perceived by the potential user, recognizing that evidence may or may not be valuable to the end user based on local circumstances and priorities. Recipients are actors involved in implementation who may be affected by and influence the implementation of evidence. Context characterizes the circumstances in which knowledge and innovation uptake occurs, consisting of multiple factors at the micro, meso, and macro levels. Finally, integral to this framework is facilitation as the active mechanism by which uptake and implementation of evidence occurs, making it an ideal and appropriate fit for this study.

All research activities for this study will be conducted in 9 children's hospitals that participate in both the SHARPS Collaborative and NSQIP-P. Our participating hospitals are geographically dispersed and (like most children's hospitals) are located in urban settings. SHARPS Collaborative hospitals feature active ASPs operated by dedicated pharmacists and physician leaders. Clinicians (MD/DO or PharmD) overseeing ASPs and surgical champions in participating hospitals will implement the proposed strategies and collect implementation outcomes that quantify the extent to which the test strategies are successfully deployed in the hospital. The daily work of these individuals to improve antibiotic use includes frequent interaction with surgical specialties that perform clean and clean-contaminated surgeries. Implementing our proposed strategies via established ASP clinicians and a surgical leader (rather than, for example, directly by a member of the research team) will leverage existing relationships between these clinicians and their associated surgical teams, creating a more realistic circumstance under which new ASP strategies are implemented. This approach will provide better insight into the feasibility of implementing these strategies in a sustainable way in the future. In addition to being SHARPS Collaborative hospitals, our participating hospitals will also be NSQIP-P hospitals, each with a full-time, trained dedicated data abstractor collecting data on surgeries and surgical outcomes.

The investigators will compare the efficacy of the two strategies designed to reduce unnecessary postoperative antibiotic prophylaxis, using a cross-sectional stepped-wedge design. The investigators have identified 9 Children's Hospitals from across the US to participate in the study. Each of the 9 hospitals will be randomized into one of 3 clusters (cluster size = 3). All hospitals will begin with the control intervention-implementation of order set review and modification-at time 0. Each Step will last 6 months. Prior to the beginning of Step 1, Cluster 1 hospitals will receive the experimental intervention -order set review and modification plus facilitation. Just prior to steps 1, 2 and 3, the ASP teams will receive a 2-day in-person workshop led by the implementation scientist (Co-I Dr. McKay) and PI Dr. Newland, covering the specific facilitation strategies to be utilized. Every 6 months, an additional cluster will initiate the experimental condition (Steps 2 and 3). The amount of time each cluster will receive the experimental condition will be 30 months (Cluster 1), 24 months (Cluster 2), and 18 months (Cluster 3). Monthly study webinars will occur with all sites in step 0. During steps 1 and 2, sites in the experimental arm will have a monthly webinar separate from the group still in the control arm. By step 3 all sites will be a part of the same monthly webinar.

ELIGIBILITY:
Inclusion Criteria:

1. Surgeries performed at the Children's Hospitals included in the study and are collected by NSQIP-P.
2. Clean and clean-contaminated surgical procedures within the following specialties that are included in NSQIP-P:

General Surgery, Neurosurgery, Orthopedics, Otolaryngology, Plastic Surgery, Otolaryngology, and Urology

Exclusion Criteria:

1. Children undergoing clean or clean-contaminated procedures that are not collected by NSQIP-P data abstractors.

Ages: 0 Days to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39363 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of clean and clean-contaminated cases in children receiving post-operative antibiotic prophylaxis. | 3 years
  Clean and clean-contaminated surgical cases in children will be assessed for whether they are receiving post operative prophylaxis utilizing the Pediatric National Surgical Quality Improvement Project (NSQIP) database. A percentage will be determined with the numerator being total number of clean and clean-contaminated cases receiving post operative surgical prophylaxis and the denominator will be total number of clean and clean-contaminated cases.

SECONDARY OUTCOMES:
Rate of Surgical Site Infections (SSI) in clean and clean-contaminated cases | 3 years
  Among the captured clean and clean-contaminated cases utilized in the primary outcome, the SSI rate per 100 cases will be determined in patients both receiving and not receiving post-operative antibiotic prophylaxis
Rate of Clostridioides difficile infections (CDI) in clean and clean-contaminated cases | 3 years
  Among the captured clean and clean-contaminated cases utilized in the primary outcome, the CDI rate per 100 cases will be determined in patients both receiving and not receiving post-operative antibiotic prophylaxis

OTHER OUTCOMES:
Implementation Outcome: Acceptability of the Interventions | 3 years
  A validated 4 question survey will be used to assess the acceptability of each intervention.
Implementation Outcome: Feasibility of the Interventions | 3 years
  A validated 4 question survey will be used to assess the feasibility of each intervention.
Implementation Outcome: Appropriateness of the Interventions | 3 years
  A validated 4 question survey will be used to assess the appropriateness of each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jason G Newland, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- United States (10):
  - Johns Hopkins University School of Medicine / Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Harvard Medical School / Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan / CS Mott Children's Hospital, Ann Arbor, Michigan
  - University of Missouri - Kansas City / The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University in St. Louis / St. Louis Children's Hospital, St Louis, Missouri
  - The Ohio State University College of Medicine / Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University / Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas
  - University of Utah / Primary Children's Hospital, Salt Lake City, Utah
  - University of Washington / Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Logan LK, Renschler JP, Gandra S, Weinstein RA, Laxminarayan R; Centers for Disease Control; Prevention Epicenters Program. Carbapenem-Resistant Enterobacteriaceae in Children, United States, 1999-2012. Emerg Infect Dis. 2015 Nov;21(11):2014-21. doi: 10.3201/eid2111.150548. PMID 26486124
- [Background] Logan LK, Braykov NP, Weinstein RA, Laxminarayan R; CDC Epicenters Prevention Program. Extended-Spectrum beta-Lactamase-Producing and Third-Generation Cephalosporin-Resistant Enterobacteriaceae in Children: Trends in the United States, 1999-2011. J Pediatric Infect Dis Soc. 2014 Dec;3(4):320-8. doi: 10.1093/jpids/piu010. Epub 2014 Mar 19. PMID 26625452
- [Background] Logan LK, Gandra S, Mandal S, Klein EY, Levinson J, Weinstein RA, Laxminarayan R; Prevention Epicenters Program, US Centers for Disease Control and Prevention. Multidrug- and Carbapenem-Resistant Pseudomonas aeruginosa in Children, United States, 1999-2012. J Pediatric Infect Dis Soc. 2017 Nov 24;6(4):352-359. doi: 10.1093/jpids/piw064. PMID 27856730
- [Background] Herigon JC, Hersh AL, Gerber JS, Zaoutis TE, Newland JG. Antibiotic management of Staphylococcus aureus infections in US children's hospitals, 1999-2008. Pediatrics. 2010 Jun;125(6):e1294-300. doi: 10.1542/peds.2009-2867. Epub 2010 May 17. PMID 20478934
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Sandora TJ, Fung M, Melvin P, Graham DA, Rangel SJ. National Variability and Appropriateness of Surgical Antibiotic Prophylaxis in US Children's Hospitals. JAMA Pediatr. 2016 Jun 1;170(6):570-6. doi: 10.1001/jamapediatrics.2016.0019. PMID 27088649
- [Background] Harvey G, Kitson A. PARIHS revisited: from heuristic to integrated framework for the successful implementation of knowledge into practice. Implement Sci. 2016 Mar 10;11:33. doi: 10.1186/s13012-016-0398-2. PMID 27013464
- [Background] Kitson AL, Rycroft-Malone J, Harvey G, McCormack B, Seers K, Titchen A. Evaluating the successful implementation of evidence into practice using the PARiHS framework: theoretical and practical challenges. Implement Sci. 2008 Jan 7;3:1. doi: 10.1186/1748-5908-3-1. PMID 18179688
- [Background] Burnham JP, Olsen MA, Kollef MH. Re-estimating annual deaths due to multidrug-resistant organism infections. Infect Control Hosp Epidemiol. 2019 Jan;40(1):112-113. doi: 10.1017/ice.2018.304. Epub 2018 Nov 22. No abstract available. PMID 30463634
- [Background] Rycroft-Malone J, Seers K, Chandler J, Hawkes CA, Crichton N, Allen C, Bullock I, Strunin L. The role of evidence, context, and facilitation in an implementation trial: implications for the development of the PARIHS framework. Implement Sci. 2013 Mar 9;8:28. doi: 10.1186/1748-5908-8-28. PMID 23497438
- [Background] Helfrich CD, Damschroder LJ, Hagedorn HJ, Daggett GS, Sahay A, Ritchie M, Damush T, Guihan M, Ullrich PM, Stetler CB. A critical synthesis of literature on the promoting action on research implementation in health services (PARIHS) framework. Implement Sci. 2010 Oct 25;5:82. doi: 10.1186/1748-5908-5-82. PMID 20973988
- [Background] Liu J, Colditz GA. Optimal design of longitudinal data analysis using generalized estimating equation models. Biom J. 2017 Mar;59(2):315-330. doi: 10.1002/bimj.201600107. Epub 2016 Nov 23. PMID 27878852
- [Background] Liu J, Colditz GA. Relative efficiency of unequal versus equal cluster sizes in cluster randomized trials using generalized estimating equation models. Biom J. 2018 May;60(3):616-638. doi: 10.1002/bimj.201600262. Epub 2018 Mar 25. PMID 29577363
- [Derived] McKay V, Malone S, Tetteh E, Saito J, Rangel S, Bono K, Tao J, Liu J, Obeng H, Atkinson A, Newland JG. Facilitation as an effective strategy to reduce excessive antibiotic prophylaxis in Children's hospitals: A stepped-wedge cluster randomized controlled trial. Implement Sci. 2025 Oct 21;20(1):45. doi: 10.1186/s13012-025-01455-2. PMID 41121325
- [Derived] McKay V, Malone S, Tetteh E, Saito J, Rangel S, Bono K, Tao J, Liu J, Obeng H, Atkinson A, Newland J. Facilitation as an effective strategy to reduce excessive antibiotic prophylaxis in Children's hospitals: A stepped-wedge cluster randomized controlled trial. Res Sq [Preprint]. 2025 May 30:rs.3.rs-6579066. doi: 10.21203/rs.3.rs-6579066/v1. PMID 40502788
- [Derived] Malone S, Bono K, Saito JM, Rangel S, Liu J, Newland JG, McKay V. Evaluating a virtual facilitation workshop with antimicrobial stewardship teams within a cluster randomized stepped-wedge trial. BMC Health Serv Res. 2024 Oct 21;24(1):1263. doi: 10.1186/s12913-024-11714-5. PMID 39434072
- [Derived] Malone S, McKay VR, Krucylak C, Powell BJ, Liu J, Terrill C, Saito JM, Rangel SJ, Newland JG. A cluster randomized stepped-wedge trial to de-implement unnecessary post-operative antibiotics in children: the optimizing perioperative antibiotic in children (OPerAtiC) trial. Implement Sci. 2021 Mar 19;16(1):29. doi: 10.1186/s13012-021-01096-1. PMID 33741048
- See also: SHARPS Collaborative Website — http://pediatrics.wustl.edu/sharps
- See also: NSQIP-P Website — https://www.facs.org/quality-programs/childrens-surgery/pediatric
- See also: American Academy of Pediatrics Choosing Wisely- Infectious Diseases — https://www.choosingwisely.org/societies/american-academy-of-pediatrics-committee-on-infectious-diseases-and-the-pediatric-infectious-diseases-society

DOCUMENTS (1):
  • Informed Consent Form (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT04366440/ICF_000.pdf